CLINICAL TRIAL: NCT03996798
Title: Disability Case Manager: Full Member of the Revalidation Team
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PXL University College (Other)
Collaborators: Jessa Hospital (Other); Revalidatie & MS Centrum Overpelt (Other); RIZIV (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PXL_WeerWerk
Record Dates: First submitted 2019-06-04; First posted 2019-06-25 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Vocational Rehabilitation
Keywords: vocational rehabilitation; back-to-work; social participation; disability case manager

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jessa Hospital, Herk-de-Stad (Experimental): "Back to Work" methodology: a revalidation trajectory with standard revalidation therapy in combination with an early focus on "back to work", using a "Disability Case Manager"
  Interventions: Other: Disability Case Manager
- Revalidation and MS Clinic Overpelt (No Intervention): Standard revalidation therapy without explicit focus on "back to work"

INTERVENTIONS:
Other: Disability Case Manager — The DCM will act as key figure between the patient, the multidisciplinary team of the revalidation centre, the employers and other back-to-work services in order to increase vocational reintegration after an incident which caused a handicap or chronic disease.
  Arms: Jessa Hospital, Herk-de-Stad

SUMMARY:
The first 4-6 months after an incident which caused a handicap or chronic disease, it is important to involve and motivate patients to return to work. After this period, there is a major decrease on successful vocational reintegration. To facilitate vocational rehabilitation a Disability Case Manager (DCM) may play a major role. The DCM will act as key figure between the patient, the multidisciplinary team of the revalidation centre, the employers and other back-to-work services. There is need to provide evidence on the value of this program. The aim of this study is to test the added value of including a DCM in the classic revalidation trajectory, who will focus on early vocational and/or social rehabilitation.

DETAILED DESCRIPTION:
12.5% of the population is confronted with a handicap or chronic disease which complicates quality of life, including the professional activities. 58% of this group is unemployed or inactive. The first 4-6 months after an incident which caused a handicap or chronic disease, it is important to involve and motivate patients to return to work. After this period, there is a major decrease on successful vocational reintegration. After 1-year unemployment, vocational reintegration decreases to 20%, which means an early intervention is recommended.

The classic rehabilitation trajectory is for the greater part directed at regaining patient's independence concerning daily activities, housing conditions, hobbies and its family. Revalidation is not (or only in the end) focused on back to work.

The revalidation centre Sint-Ursula, Jessa Hospital, Hasselt developed an interdisciplinary methodology 'Back-To-Work', which included an early focus on vocational and/or social rehabilitation using a 'Disability Case Manager (DCM)'. The DCM act as key figure between the patient, the multidisciplinary team of the revalidation centre, the employers and other back-to-work services to facilitate return to work.

The program is initiated by an interdisciplinary screening at time of hospitalisation. Together with the patient, there can be chosen for two revalidation pathways: 1/ focus on vocational rehabilitation; or 2/ focus on social participation. The labour pathway includes the matching of the persons characteristics and capacity with the requirements of the job, followed by a task-oriented vocational training; the social participation pathway consists of guidance to alternative daytime activities combined with psychological support in coping and acceptance. The combination of these components with the focus on vocational rehabilitation and social participation is new in rehabilitation services.

Previous research, testing the involvement of a DCM, showed empirically better results, with more patients going back to work or choosing an alternative job. Even when back to work was eventually not possible, those patients reported a better quality of life.

This project aims at a scientifically validation of the 'Back-To-Work' methodology and the role of DCM. Patients with complex neuro-locomotoric conditions and amputations, aged between 18-62 years, will be asked to participate in a controlled, longitudinal study, receiving either a revalidation therapy including the experimental 'Back-to-work' methodology (Jessa hospital, campus Sint-Ursula) or a standard revalidation therapy (Revalidation & MS Clinic Overpelt, control group). At the start of rehabilitation, at the end of rehabilitation and 6 months after rehabilitation, data for qualitative and quantitative analysis is gathered.

ELIGIBILITY:
Inclusion Criteria:

* Complex neuro-motoric conditions
* Age between 18-62 year
* Working
* Persons belonging to the National Institute for Health and Disability Insurance (NIHDI) target group

Exclusion Criteria:

* Comatose patients
* Retired patients
* Students
* Persons who not belong to the NIHDI target group

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life: Short Form 36 questionnaire | pre (at moment of inclusion), post (at the end of the revalidation period, on average after 6 months) and follow-up (6 months after revalidation)
  Short Form 36 questionnaire. This questionnaire includes 11 questions with different scale ranges and contents.
Change in mental functioning: depressive feelings, anxiety and stress | pre (at moment of inclusion), post (at the end of the revalidation period, on average after 6 months) and follow-up (6 months after revalidation)
  Depression, Anxiety and Stress scale 21 questionnaire. Scale ranges from 0 to 3 (0 = never applicable, 1 = sometimes applicable, 2 = often applicable, 3 = certainly applicable). The lower values represent a better outcome.
Change in functional status | pre (at moment of inclusion), post (at the end of the revalidation period, on average after 6 months) and follow-up (6 months after revalidation)
  Barthel Activities of Daily Living (ADL) index. Scale ranges from 0 to 2 or 3, each topic (feeding, bathing, grooming, dressing, bowels, bladder, toilet use, transfers (bed to chair and back), mobility and stairs) has its own scale content. The higher values represent a better outcome.
Change in participation | pre (at moment of inclusion), post (at the end of the revalidation period, on average after 6 months) and follow-up (6 months after revalidation)
  Nottingham ADL index. Scale ranges from 0 to 3 (0 = patient can not execute the activity, 1 = patient can execute the activity with help, 2 = patient can execute the activity, but it is still difficult, 3 = patient can execute the activity easily). The higher values represent a better outcome.
Change in work status (questionnaire) | pre (at moment of inclusion), post (at the end of the revalidation period, on average after 6 months) and follow-up (6 months after revalidation)
  Follow up of current working status. Scales ranges from 0 to 7 (0 = no work, 1 = retirement, 2 = volunteer work, 3 = still in support of re-employment, 4 = half time other work, 5 = other work, 6 = half time same work, 7 = same work)

SECONDARY OUTCOMES:
Change in coping | pre (at moment of inclusion), post (at the end of the revalidation period, on average after 6 months) and follow-up (6 months after revalidation)
  Coping Inventory of Stressful Situations (CISS), the Utrecht Coping list. Scales ranges from 1 to 5 (1 = not at all, 5 = very strong).
Change in self-effectiveness | pre (at moment of inclusion), post (at the end of the revalidation period, on average after 6 months) and follow-up (6 months after revalidation)
  Dutch General Self-Efficacy Scale (SES). Scale ranges from 1 to 4 (1 = completely incorrect, hardly correct, slightly correct, completely correct).
Expectations concerning back-to-work | pre (at moment of inclusion)
  Worker Role Interview. This interview includes open questions about the consequences of the incident, the current and previous employments and back to work after the revalidation.
Change in satisfaction with revalidation traject | post (at the end of the revalidation period, on average after 6 months) and follow-up (6 months after revalidation)
  Questionnaire. The scales range from 0 to 3 or 1 to 5. (0-3: 0 = strongly disagree, 1 = disagree, 2 = agree, 3 = strongly agree; 1-5: 1 = not at all, 2 = to some extent, 3 = to a reasonable extent, 4 = to a large extent, 5 = to a very large extent). The higher values represent a better outcome.
Change in expectations concerning back-to-work | pre (at moment of inclusion), post (at the end of the revalidation period, on average after 6 months) and follow-up (6 months after revalidation)
  Questionnaire. The scale ranges from 1 to 5 (1 = not at all, 2 = to some extent, 3 = to a reasonable extent, 4 = to a large extent, 5 = to a very large extent). The higher values represent a better outcome.
Satisfaction with revalidation traject and back-to-work focus: Semi-structured interview | follow-up (6 months after revalidation)
  Semi-structured interview. This interview includes open questions.

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Spooren, PhD, Principal Investigator — PXL University College
Locations (2):
- Belgium (2):
  - Jessa Hospital, Campus Sint-Ursula, Hasselt, Limburg
  - Revalidation & MS Clinic Overpelt, Overpelt, Limburg

IPD SHARING:
Plan to Share IPD: No